CLINICAL TRIAL: NCT04358744
Title: The Real World Study of Children With Autism Spectrum Disorder in China
Brief Title: The Real World Study of Autism Spectrum Disorder in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-20-005
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood and stool samples are retained in Xinhua
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators conduct the real world study to explore mechanisms of autism based on multi-modal data.

DETAILED DESCRIPTION:
Children with autism spectrum disorder registered in Xinhua Hospital are measured in aspects of behavioural accessment, genetic test, blood lab test, gut microbiome and neuroimaging including structural and functional magnetic resonance imaging (MRI), functional near - infrared spectroscopy(f-NIRS), electroencephalography and eye movement. The investigators conduct the real world study to explore mechanisms of autism based on the multi-modal data.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with autism spectrum disorder
* registered in Xinhua hospital
* written informed consent provided

Exclusion Criteria:

* NA

Ages: 18 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with autism spectrum disorder have registered in Xinhua hospital and provided written informed consent from themselves and/or their legal guardians.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2019-04-13 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Behaviour assessment | The baseline and 3 months
  The behaviour development of participants includes intellectual/developmental quotient, syptoms severity, comorbidity, etc.

OTHER OUTCOMES:
Genetic characteristics | The baseline
  Genome wide association study from blood sample
Blood test | The baseline and 3 months
  Retained blood samples tested in immunomics, metabonomics, etc
Blood test | The baseline and 6 months
  Retained blood samples tested in immunomics, metabonomics, etc
Blood test | The baseline and 12 months
  Retained blood samples tested in immunomics, metabonomics, etc
Gut mircobiome | The baseline and 1 months
  Retained stool samples tested in metabonomics, genomics, etc
Gut mircobiome | The baseline and 3 months
  Retained stool samples tested in metabonomics, genomics, etc
Gut mircobiome | The baseline and 6 months
  Retained stool samples tested in metabonomics, genomics, etc
Gut mircobiome | The baseline and 12 months
  Retained stool samples tested in metabonomics, genomics, etc
Head Magnetic Resonance Imaging (Head MRI) | The baseline and 3 months
  Head MRI is used to detect the structure and function of the brain.
Head Magnetic Resonance Imaging (Head MRI) | The baseline and 12 months
  Head MRI is used to detect the structure and function of the brain.
Functional near - infrared spectroscopy(f-NIRS) | The baseline and 3 months
  Head fNIRs is a non-invasive, non-ionizing method for measuring and imaging the functional hemodynamic response to brain activity. It measures changes in hemoglobin (Hb) concentrations within the brain by means of the characteristic absorption spectra of Hb in the near-infrared range.
Functional near - infrared spectroscopy(f-NIRS) | The baseline and 6 months
  Head fNIRs is a non-invasive, non-ionizing method for measuring and imaging the functional hemodynamic response to brain activity. It measures changes in hemoglobin (Hb) concentrations within the brain by means of the characteristic absorption spectra of Hb in the near-infrared range.
Functional near - infrared spectroscopy(f-NIRS) | The baseline and 12 months
  Head fNIRs is a non-invasive, non-ionizing method for measuring and imaging the functional hemodynamic response to brain activity. It measures changes in hemoglobin (Hb) concentrations within the brain by means of the characteristic absorption spectra of Hb in the near-infrared range.
Multichannel Electroencephalography signals | The baseline and 3 months
  The latency and amplitude measured by electroencephalogram can reflect the connectivity between brain regions.
Multichannel Electroencephalography signals | The baseline and 6 months
  The latency and amplitude measured by electroencephalogram can reflect the connectivity between brain regions.
Multichannel Electroencephalography signals | The baseline and 12 months
  The latency and amplitude measured by electroencephalogram can reflect the connectivity between brain regions.
Eye movements | The baseline and 3 months
  Variables measured by eye movements represent cognition.
Eye movements | The baseline and 6 months
  Variables measured by eye movements represent cognition.
Eye movements | The baseline and 12 months
  Variables measured by eye movements represent cognition.
Behaviour assessment | The baseline and 6 months
  The behaviour development of participants includes intellectual/developmental quotient, syptoms severity, comorbidity, etc.
Behaviour assessment | The baseline and 12 months
  The behaviour development of participants includes intellectual/developmental quotient, syptoms severity, comorbidity, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, doctor, Principal Investigator — Xinhua hospital Affilated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- ShanghaiXinhua, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No